CLINICAL TRIAL: NCT07044895
Title: Evaluation of Diode Laser Photocoagulation With Immediate Implant Placement in the Maxillary Esthetic Zone
Brief Title: Diode Laser Photocoagulation With Immediate Implant Placement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Lecturer of Dental Public Health and biostatistical consultanat, Alexandria University
Organization: Alexandria University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-H-0167-D-M-0754
Record Dates: First submitted 2025-06-22; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Tooth Extraction; Immediate Dental Implant; Photocoagulation; Maxillary Esthetic Zone
MeSH Terms: interventions — Lasers, Semiconductor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immediate implant with photocoagulation (Experimental)
  Interventions: Other: Diode laser and Immediate implant

INTERVENTIONS:
Other: Diode laser and Immediate implant — patients with non-restorable teeth in the maxillary esthetic zone will be included in this prospective single-arm study. The non-restorable tooth will be atraumatically extracted and immediate implant placement will be placed. The extraction socket will be sealed with diode laser photocoagulation and customized healing abutments fabrication.

SUMMARY:
Placement of an immediate implant is becoming popular because of its potential in minimizing the treatment time and enhancing the patient comfort and esthetic outcomes. It is crucial to maintain adequate thickness of labial bone with the establishment of a stable and healthy gingival seal around the implant abutment to prevent the invasion of bacteria and peri-implant inflammation. Diode lasers have been developed as a promising tool in dentistry, providing a precise manipulation and photocoagulation effect that may have a positive influence on both bone remodeling and soft tissue healing. This study aims to evaluate the effectiveness of the utilization of diode laser photocoagulation with immediate implant placement and customized healing abutment in the maxillary esthetic zone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-restorable maxillary teeth in the aesthetic zone are indicated for extraction and subsequent immediate implant placement, including those with:
* A severely carious tooth that cannot be restored.
* Pulpal necrosis or irreversible pulpitis that is not amenable to endodontics.
* Periodontally involved teeth with grade 2 mobility or above.
* Teeth with root caries that can't be restored.
* Patients with an extraction socket Type I.
* A good standard of oral hygiene.

Exclusion Criteria:

* Patients with extraction socket Type II or III, with buccal plate defects.
* Absence of at least 2 mm of bone apical to the extraction socket
* tooth ankylosis.
* Patients with deciduous teeth.
* Heavy smokers.
* Systemic conditions
* History of oral or intravenous bisphosphonate therapy or any treatments with other medications that may interfere with bone metabolism within the past 12 months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Change in pain socres | at 7, 14, and 21 days
  Pain will be evaluated, using visual analogue scale (VAS) as follows:
  (0-1= None, 2-4= Mild, 5-7= Moderate, 8-10= Severe)
Change in wound healing | at 7, 14, and 21 days
  The wound healing will be assessed based on Landry Wound Healing Index. The Landry Index uses a numerical score based on the assessment of four given parameters (Erythema, Edema, Wound Margin Adaptation, and Presence of Exudate). Each parameter is given a score depending on its severity, and the total score determine an overall evaluation of wound healing
Change in implant stability | baseline and 6 months
  The base line primary Implant Stability Quotient (ISQ) will be measured during the operative stage, while the secondary stability quotient will be measured 6-months post-operative during the prosthetic phase preparation.

SECONDARY OUTCOMES:
Change in Crestal Alveolar Process width | baseline and 6 months
  The width of the crestal alveolar process will be assessed by determination of the dimensional changes of Bucco-palatal ridge in the 6 months' scan
Change in labial bone thickness | baseline and 6 months
  The overall persistence of the labial plate of bone after the atraumatic extraction and immediate implant placement will be evaluated by the assessment of the thickness labial plate of bone in the scan performed after 6 months and comparing it with the preoperative CBCT record. The distance will be measured from the root surface to the outer buccal bone surface in the preoperative CBCT record. Measurements will be performed on the cross-sectional cut of the CBCT at three levels; crestal labial thickness, middle labial thickness, and apical labial thickness.
Change in esthetic of soft tissue | at 1 month
  The pink esthetic score (PES) introduced by Furhauser et al will be used for evaluation of the esthetic outcome of soft tissue surrounding single crowns supported by implant in the esthetic zone. The PES consists of seven factors each one is given a score of 2, 1, or 0, and a total score will be ranging between 0 and 14

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry clinics, Beirut Arab University, Beirut, Lebanon